CLINICAL TRIAL: NCT05637515
Title: A Multicenter, Randomized, Blinded, Parallel Group, Interchangeability Study in Moderate to Severe Chronic Plaque Psoriasis Evaluating Pharmacokinetics, Efficacy, Safety, and Immunogenicity Between Subjects Receiving Humira® Pre Filled Syringe (40 mg) Continuously and Subjects Undergoing Repeated Switches Between Humira® Pre Filled Syringe (40 mg) and Hulio Pre-filled Syringe (40 mg)
Brief Title: Hulio Interchangeability to Humira®, Comparing Pharmacokinetics, Efficacy, Safety and Immunogenicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocon Biologics Inc. (Industry)
Collaborators: Mylan Inc. (Industry); MEDA Pharma GmbH & Co. KG (Industry); IQVIA Pvt. Ltd (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADA-IJZ-3001; 2021-006015-29 (EudraCT Number)
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Moderate Chronic Plaque Psoriasis; Severe Chronic Plaque Psoriasis
Keywords: adalimumab; pharmacokinetics; plaque psoriasis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Humira continuously (Active Comparator): Subjects receive Humira continuously both during Run-in period and Randomized interchangeable treatment period.
  Run-in Period:
  Subjects will receive Humira (initial dose of 80 mg [2 × 40 mg]; Day 1 administered subcutaneously (SC), followed by 40 mg SC given every other week starting 1 week after the initial dose (last dose at Week 10).
  Randomized interchangeable treatment period:
  Subjects continue to receive Humira (40 mg every other week) until Week 26
  Interventions: Biological: Humira 40 MG in Prefilled Syringe
- Repeated switches Humira - Hulio (Experimental): Subjects will receive Humira in Run-in period & undergo repeated switches between Humira Hulio during randomized interchangeable treatment period
  Randomized interchangeable treatment period:
  * Subjects undergo repeated switches between Humira and Hulio between week 12 to week 26.
  * Hulio (40 mg every other week) at Week 12 and Week 14
  * Humira (40 mg every other week) at Week 16 and Week 18, and
  * Hulio (40 mg every other week) at Week 20, Week 22, Week 24 and Week 26.
  Interventions: Biological: Hulio 40 MG in Prefilled Syringe / Humira 40 MG in Prefilled Syringe

INTERVENTIONS:
Biological: Humira 40 MG in Prefilled Syringe — Humira (40 mg every other week)
  Arms: Humira continuously
Biological: Hulio 40 MG in Prefilled Syringe / Humira 40 MG in Prefilled Syringe — • Subjects will receive Humira (initial dose of 80 mg [2 × 40 mg]; Day 1 administered subcutaneously (SC), followed by 40 mg SC given every other week starting 1 week after the initial dose (last dose at Week 10).
  Hulio (40 mg every other week) at Week 12 and Week 14
  * Humira (40 mg every other week) at Week 16 and Week 18, and
  * Hulio (40 mg every other week) at Week 20, Week 22, Week 24 and Week 26.
  Arms: Repeated switches Humira - Hulio

SUMMARY:
Hulio is a monoclonal antibody currently approved as a biosimilar to European Union approved and United States (US)-Licensed Humira.

This is a multicenter, randomized blinded, parallel group, interchangeability study in subjects with moderate to severe chronic plaque psoriasis, undergoing repeated switches between Humira and Hulio. The study is designed to confirm the pharmacokinetic equivalence of alternating between the use of Humira and Hulio and, Humira without such alternation or switch, in accordance with the US Food and Drug Administration Guidance for Industry, Considerations in Demonstrating Interchangeability with a Reference Product.

The study will also assess safety, efficacy and immunogenicity between these two groups.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Able to understand and voluntarily provide written informed consent to participate in the study
2. Aged 18 to 75 years, inclusive, at the time of Screening
3. Has moderate to severe chronic plaque psoriasis for at least 6 months prior to screening and that has involved body surface area ≥10%, PASI ≥12, and static Physicians Global Assessment (sPGA) ≥3 (moderate) at Screening and at Baseline
4. Has stable disease for at least 2 months (i.e., without significant changes as defined by the principal investigator [PI] or designee)
5. Is a candidate for systemic therapy or phototherapy
6. Has a previous failure, inadequate response, intolerance, or contraindication to at least 1 conventional antipsoriatic systemic therapy, including methotrexate, cyclosporine, psoralen plus ultraviolet light A (PUVA), and ultraviolet light B (UVB)
7. Willing to follow the contraception requirement, based on the childbearing potential.

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

1. Has been diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (e.g., eczema), or other systemic autoimmune disorder/ inflammatory disease at the time of the Screening visit that would interfere with evaluations of the effect of the study treatment of psoriasis
2. Prior and concomitant medications: Has prior use of any of the medications specified in the CTP within specified time periods or will require use during the study:
3. Has received live or attenuated vaccines during the 4 weeks prior to Screening or has the intention of receiving a live or attenuated vaccine at any time during the study
4. Other medical conditions: Known chronic or relevant acute TB
5. Has an underlying condition (including, but not limited to, metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal) which, in the opinion of the PI or designee, significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy
6. Has a planned surgical intervention during the duration of the study and which, in the opinion of the PI or designee, will put the subject at further risk or hinder the subject's ability to maintain compliance with study treatment and the visit schedule
7. Has any active and serious infection or history of infections
8. Is positive for human immunodeficiency virus (HIV), hepatitis C virus antibody, or hepatitis B surface antigen (HbsAg) or is positive for hepatitis B core antibody (HbcAb) at Screening
9. Has laboratory abnormalities, including but not limited to clinically significant hematological abnormalities, that, in the opinion of the PI or designee, could cause this study to be detrimental to the subject. The subjects should be excluded if they have the following laboratory abnormalities

   1. Hemoglobin <9 g/dL
   2. Platelet count <100 000/mm3
   3. White blood cell count <3000 cells/mm3
   4. Aspartate aminotransferase and/or alanine aminotransferase that is persistently ≥2.5 × the upper limit of normal. (Persistently indicates elevated transaminases, at least on two separate occasions)
   5. Creatinine clearance <50 mL/min (Cockcroft Gault formula)
10. Has severe progressive or uncontrolled, clinically significant disease that in the judgment of the PI or designee renders the subject unsuitable for the study
11. Has moderate to severe heart failure (New York Heart Association [NYHA] Class III/IV)
12. Has a history of hypersensitivity to the active substance or to any of the excipients of Humira or Hulio
13. Is pregnant or nursing (lactating) woman
14. Has evidence (as assessed by the PI or designee using good clinical judgment) of alcohol or drug abuse or dependency up to 5 years prior to Screening
15. Is unable to follow study instructions and comply with the protocol in the opinion of the PI or designee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- Bulgaria (10):
  - Site 407 - Medical Centre "Asklepii", OOD, Dupnitsa
  - Site 409 - Medical center Medconsult Pleven OOD, Pleven
  - Site 403 - MC Rusemed ltd., Rousse
  - Site 406 - Medical Center Unimed Eood, Sevlievo
  - Site 401 - Ambulatory for Specialized Medical Help - skin and venereal diseases, Sofia
  - Site 402 - DCC "Alexandrovska", EOOD, Sofia
  - Site 404 - DCC Focus 5 - MEOH OOD, Sofia
  - Site 405 - Medical Center Hera EOOD, Sofia
  - Site 408 - DCC "Alexandrovska", EOOD, Sofia
  - Site 410 - DCC XXVIII, Sofia
- Czechia (4):
  - Site 304 - CCR Ostrava s.r.o., Ostrava
  - Site 303 - CCR Czech, a.s., Pardubice
  - Site 301 - Kozni Ambulance Fialova s.r.o., Prague
  - Site 302 - CLINTRIAL s.r.o., Prague
- Estonia (4):
  - Site 203 - North Estonia Medical Centre Foundation, Talinn
  - Site 201 - Tartu University Hospital, Tartu
  - Site 204 - Clinical Research Centre, Tartu
  - Site 205 - OÜ Innomedica, Tartu
- Poland (18):
  - Site 104 - Clinic Med Daniluk, Nowak Spółka Jawna, Bialystok
  - Site 111 - SPECDERM POZNANSKA, Bialystok
  - Site 103 - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Site 101 - Centrum Kliniczno - Badawcze J. Brzezicki, B. Górnikiewicz-Brzezicka Lekarze Spółka Partnerska, Elblag
  - Site 109 - Centrum Badan Klinicznych P.I. House Sp. z o.o., Gdansk
  - Site 112 - CENTRUM MEDYCZNE ALL-MED, Krakow
  - Site 116 - FutureMeds Krakow, Krakow
  - Site 106 - ETG Lodz, Lodz
  - Site 108 - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - Site 115 - ETG Lublin, Lublin
  - Site 113 - ai centrum medyczne sp. z o.o. sp.k., Poznan
  - Site 120 - Twoja Przychodnia PCM, Poznan
  - Site 118 - ETG Siedlce, Siedlce
  - Site 114 - ETG Skierniewice, Skierniewice
  - Site 105 - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Site 107 - MICS Centrum Medyczne Warszawa, Warsaw
  - Site 110 - Clinical Research Group Sp. z o.o., Warsaw
  - Site 117 - MCM POLIMEDICA, Warsaw

REFERENCES:
- [Derived] Deodhar S, Loganathan S, Kadadanamari Subbarama Reddy R, Ranganna GM, Liu S, Hummel MA, Daniluk S, Hanczewska A, Vekovska K, Zegadlo-Mylik M, Pulka G, -Holz EW. Multiple Switches Between Adalimumab-fkjp and Reference Adalimumab in Moderate-to-Severe Chronic Plaque Psoriasis: A Multicenter, Double-Blind, Parallel Group, Randomized Clinical Trial for Interchangeability. Adv Ther. 2025 Aug;42(8):3795-3809. doi: 10.1007/s12325-025-03240-5. Epub 2025 Jun 10. PMID 40493334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 374 subjects were randomized into the randomized interchangeable treatment period which comprised of two groups, Group 1 and Group 2. Subjects in Group 1 (N=193), continued to receive Humira (40 mg every other week) until Week 26/Visit 14; While subjects in Group 2 (N=181), underwent multiple switches until Week 26/Visit 14: Hulio (40 mg every other week) for 4 weeks, Humira (40 mg every other week) for 4 weeks, and Hulio (40 mg every other week) for 8 weeks.
Groups:
- Group 1 :- Humira Continuously: Subjects received Humira continuously during both periods:
  Run-in Period: Initial Humira 80 mg dose (two 40 mg doses) on Day 1, followed by 40 mg SC every other week from Week 1 to Week 10.
  Randomized Interchangeable Treatment Period: 40 mg SC every other week until Week 26/Visit 14.
- Group 2:- Repeated Switches Humira - Hulio: Subjects switched between Humira and Hulio:
  Run-in Period: Humira 80 mg on Day 1, then 40 mg SC every other week until Week 10.
  Randomized Period: Switched treatments until Week 26:
  1. Hulio 40 mg every other week for 4 weeks.
  2. Humira 40 mg every other week for 4 weeks.
  3. Hulio 40 mg every other week for 8 weeks. Randomization was based on Week 12 PASI response.
Period: Overall Study
Arm/Group | Group 1 :- Humira Continuously | Group 2:- Repeated Switches Humira - Hulio
Started | 193 | 181
Completed | 176 | 164
Not Completed | 17 | 17
Not completed — Withdrawal by Subject | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Group 2 :- Repeated Switches Humira - Hulio: Subjects switched between Humira and Hulio:
  Run-in Period: Humira 80 mg on Day 1, then 40 mg SC every other week until Week 10.
  Randomized Period: Switched treatments until Week 26:
  1. Hulio 40 mg every other week for 4 weeks.
  2. Humira 40 mg every other week for 4 weeks.
  3. Hulio 40 mg every other week for 8 weeks.
  Randomization was based on Week 12 PASI response.
- Total: Total of all reporting groups
Arm/Group | Group 1 :- Humira Continuously | Group 2 :- Repeated Switches Humira - Hulio | Total
Number analyzed (Participants) | 193 | 181 | 374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 173 | 158 | 331
  >=65 years | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (12.86) | 45.7 (13.40) | 46.0 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 69 | 130
  Male | 132 | 112 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 192 | 179 | 371
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 191 | 181 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Czechia | 32 | 30 | 62
  Poland | 112 | 100 | 212
  Bulgaria | 45 | 46 | 91
  Estonia | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoints: Pharmacokinetics (PK) - AUC
Description: AUCτ, 26-28 (Area under the adalimumab concentration-time curve [AUC] over the dosing interval of Week 26-28)
Time Frame: Week 26 - 28
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Group 1 :- Humira Continuously | Group 2:- Repeated Switches Humira - Hulio
Number analyzed (Participants) | 166 | 159
h*ug/mL | 2127.57 (1432.80) | 2357.61 (1636.09)

2. Primary Outcome: Primary Endpoints: Pharmacokinetics (PK) - Cmax
Description: Cmax, 26-28 (Maximum observed adalimumab concentration during the dosing interval Week 26-28).
Time Frame: Week 26 - 28
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Group 1 Humira Continuously: Subjects received Humira continuously during both periods:
  Run-in Period: Initial Humira 80 mg dose (two 40 mg doses) on Day 1, followed by 40 mg SC every other week from Week 1 to Week 10.
  Randomized Interchangeable Treatment Period: 40 mg SC every other week until Week 26/Visit 14.
Arm/Group | Group 1 Humira Continuously | Group 2 :- Repeated Switches Humira - Hulio
Number analyzed (Participants) | 166 | 159
ug/mL | 7.69 (4.96) | 8.46 (5.42)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: One subject in Group 2, died due to COVID-19 pneumonia. The details of adverse events leading to death
Groups:
- Group 1:- Humira Continuously: Subjects received Humira continuously during both periods:
  Run-in Period: Initial Humira 80 mg dose (two 40 mg doses) on Day 1, followed by 40 mg SC every other week from Week 1 to Week 10.
  Randomized Interchangeable Treatment Period: 40 mg SC every other week until Week 26/Visit 14.
- Group 2:- Repeated Switches Humira - Hulio: Subjects switched between Humira and Hulio:
  Run-in Period: Humira 80 mg on Day 1, then 40 mg SC every other week until Week 10.
  Randomized Period: Switched treatments until Week 26:
  1. Hulio 40 mg every other week for 4 weeks.
  2. Humira 40 mg every other week for 4 weeks.
  2. Hulio 40 mg every other week for 8 weeks. Randomization was based on Week 12 PASI response.
Arm/Group | Group 1:- Humira Continuously | Group 2:- Repeated Switches Humira - Hulio
All-Cause Mortality (participants affected / at risk) | 0/193 | 1/181
Serious Adverse Events (participants affected / at risk) | 3/193 | 3/181
Other Adverse Events (participants affected / at risk) | 66/193 | 54/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1:- Humira Continuously (N=193) | Group 2:- Repeated Switches Humira - Hulio (N=181)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1:- Humira Continuously (N=193) | Group 2:- Repeated Switches Humira - Hulio (N=181)
Nasopharyngitis (Infections and infestations) | 11 (11) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Pharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 3 (10) | 3 (4)
Injection site pain (General disorders) | 4 (6) | 1 (1)
Injection site pruritus (General disorders) | 2 (6) | 2 (4)
Injection site swelling (General disorders) | 2 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 6 (8) | 4 (6)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (5) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (3) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish or present the results of Institution. Institution and Investigator are required to submit any proposed publication or presentation to Sponsor for review at least 30 days prior to submitting any such proposed publication. Sponsor shall advise Institution and/or Investigator, as the case may be, in writing of any information contained therein which is Confidential Information (other than Study Data).

DOCUMENTS (2):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT05637515/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT05637515/SAP_001.pdf